CLINICAL TRIAL: NCT01422057
Title: Risk Prediction in Type II Diabetics With Ischemic Heart Disease by Cardiac Autonomic Function
Brief Title: Risk Prediction in Type II Diabetics With Ischemic Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Thebiosignals.com (Other)
Responsible Party: Principal Investigator, Axel Bauer, Prof. Dr. med. Axel Bauer, Thebiosignals.com
Other Study IDs: 402/2009BO2-2
Record Dates: First submitted 2011-08-09; First posted 2011-08-23 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Type-2 Diabetes Mellitus; Ischemic Heart Disease
Keywords: diabetes; coronary artery disease; ischemic heart disease; autonomic function; heart rate turbulence; deceleration capacity; severe autonomic failure
MeSH Terms: conditions — Myocardial Ischemia; Diabetes Mellitus; Coronary Artery Disease; Pure Autonomic Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to test whether cardiac autonomic dysfunction predicts is a prognostic marker in type-2 diabetics with ischemic heart disease

DETAILED DESCRIPTION:
In patients with type 2-diabetes and ischemic heart disease autonomic function might be seriously affected.

In the present study, markers of cardiac autonomic dysfunction, repolarization and respiration abnormalities will be assessed from Holter recordings and 30-minute recordings of high-resolution three dimensional ECG, non-invasive arterial blood pressure and respiratory activity.

The correlation between markers of cardiac autonomic dysfunction and markers of severity of type-2 diabetes will be assessed. Autonomic dysfunction is assumed present when both heart rate turbulence and deceleration capacity are abnormal ("severe autonomic failure"). Assessment of severity of diabetes includes levels of HbA1c and urine albumine, duration and treatment of diabetes, and diabetes related complications (nephropathy, neuropathy, retinopathy).

ELIGIBILITY:
Inclusion Criteria:

* type-2 diabetes
* coronary artery disease

Exclusion Criteria:

* age >80 years
* acute coronary syndrome
* life expectancy <1 year
* unable to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with diagnose of ischemic heart disease and type-2 diabetes are included.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-01; Primary Completion 2014-01 (Actual); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Major cardiovascular event | 2 years
  Combination of total mortality, non-fatal myocardial infarction and non-fatal stroke

SECONDARY OUTCOMES:
Cardiovascular mortality | 2 years
sudden cardiac death | 2 years
Total mortality | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Tübingen, Tübingen, Germany